CLINICAL TRIAL: NCT04570072
Title: Effect of Probiotic on Chinese Patients With Depression and Constipated Comorbidity
Brief Title: Effect of Probiotic on Comorbidity of Depression and Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Agricultural University (Other)
Collaborators: The Affiliated Nanjing Hospital of Nanjing University of Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Fazheng Ren, professor, China Agricultural University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAUDepression-02
Record Dates: First submitted 2020-09-22; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Comorbidity of Depression and Constipation
MeSH Terms: conditions — Constipation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Formula probiotic contains freeze-dried Lactobacillus paracasei, Bifidobacterium animals, Bifidobacterium longum, Bifidobacterium bifidum, and Lactobacillus plantarum, each at a dosage of 3.0 × 10^10 colony forming unit per 2g sachet.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo made with only the excipients. The placebo sachet was matched to the study probiotic products for taste, color, and size.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Patients receive the formula probiotic for consecutive 8 weeks ( one sachet per day ).
  Arms: Probiotic
Dietary Supplement: Placebo — Patients receive the placebo identical to probiotic for consecutive 8 weeks ( one sachet per day ).
  Arms: Placebo

SUMMARY:
Depressive disorder, also known as depression, is a type of mood disorder characterized by persistent low mood. The incidence of depression worldwide is about 6%. The high comorbidity rate between depression and constipation indicated the role of the gut-brain axis in depression. Growing evidence suggested that the gut microbiota plays a key role in the development of depression. Probiotics can effectively improve constipation and regulate gut microbiota, and showed potential in alleviating depression. This study investigated the effect of formula probiotic (containing Lactobacillus paracasei, Bifidobacterium animals, Bifidobacterium longum, Bifidobacterium bifidum, and Lactobacillus plantarum) on the comorbidity of depression and constipation.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index ≥ 18.5 until ≤ 29.9
* Hamilton Rating Scale for Depression (HAMD-17) score not less than 8
* Meet the ROME III criteria for functional constipation
* Agreed to intake study product during the study period
* Agreed to sign written informed consent

Exclusion Criteria:

* Use of systemic antibiotics or antimycotics medication in the 30 days prior to the study
* Investigator's uncertainty about the willingness or ability of subject to comply with the protocol requirements
* Persons with a milk protein allergy, lactose intolerance
* Pregnant or breastfeeding women
* Subject had other serious diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Change from baseline score to intervention measurements at 4 and 8 weeks
  Depressive symptoms as measured with the Hamilton Rating Scale for Depression. The score rangs from 0 to 53. The higher score means severer depressive symptoms.

SECONDARY OUTCOMES:
Patient Assessment of Constipation Symptom | changes from baseline score to intervention measurements at 4 and 8 weeks
  Constipation symptoms as measured with the Patient Assessment of Constipation Symptom. The score ranges from 0 to 48. The higher score means severer constipated symptoms.
Serum Il-1β | changes from baseline level to intervention measurements at 4 and 8 weeks
  Serum Il-1β levels before and after intervention assessed by ELISA.
Serum Il-6 | changes from baseline level to intervention measurements at 4 and 8 weeks
  Serum Il-6 levels before and after intervention assessed by ELISA.
Serum TNF-α | changes from baseline level to intervention measurements at 4 and 8 weeks
  Serum TNF-α levels before and after intervention assessed by ELISA.
Serum cortisol | changes from baseline level to intervention measurements at 4 and 8 weeks
  Serum cortisol levels before and after intervention assessed by ELISA.
Serum Brain-derived neurotrophic factor | changes from baseline level to intervention measurements at 4 and 8 weeks
  Serum Brain-derived neurotrophic factor levels before and after intervention assessed by ELISA.
Serum concentrations of tryptophan metabolites | Changes from baseline level to intervention measurements at 4 and 8 weeks
  Serum concentrations of tryptophan metabolites quantified by High-Performance Liquid Chromatography and Mass Spectrometry
Serum concentrations of bile acid | Changes from baseline level to intervention measurements at 4 and 8 weeks
  Quantification by High-Performance Liquid Chromatography and Mass Spectrometry
Fecal microbiome | Changes from baseline to intervention measurements at 4 and 8 weeks
  Fecal microbiome measured by next generation sequencing
Stool form | Change from baseline score to intervention measurements at 4 and 8 weeks
  Stool form measured with the Bristol Stool Form Scale, which classify the form of human faeces into seven types, successively named type 1 to type 7. Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicating lack of dietary fiber, and 6 and 7 indicate diarrhoea.

CONTACTS AND LOCATIONS:
Overall Officials: Fazhen Ren, PhD, Principal Investigator — China Agricultural University
Locations (1):
- The Affiliated Nanjing Hospital of Nanjing University of Chinese Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bromet E, Andrade LH, Hwang I, Sampson NA, Alonso J, de Girolamo G, de Graaf R, Demyttenaere K, Hu C, Iwata N, Karam AN, Kaur J, Kostyuchenko S, Lepine JP, Levinson D, Matschinger H, Mora ME, Browne MO, Posada-Villa J, Viana MC, Williams DR, Kessler RC. Cross-national epidemiology of DSM-IV major depressive episode. BMC Med. 2011 Jul 26;9:90. doi: 10.1186/1741-7015-9-90. PMID 21791035
- [Background] Walker EA, Katon WJ, Jemelka RP, Roy-Bryne PP. Comorbidity of gastrointestinal complaints, depression, and anxiety in the Epidemiologic Catchment Area (ECA) Study. Am J Med. 1992 Jan 24;92(1A):26S-30S. doi: 10.1016/0002-9343(92)90133-v. PMID 1531168
- [Background] Sharon G, Sampson TR, Geschwind DH, Mazmanian SK. The Central Nervous System and the Gut Microbiome. Cell. 2016 Nov 3;167(4):915-932. doi: 10.1016/j.cell.2016.10.027. PMID 27814521
- [Background] De Palma G, Blennerhassett P, Lu J, Deng Y, Park AJ, Green W, Denou E, Silva MA, Santacruz A, Sanz Y, Surette MG, Verdu EF, Collins SM, Bercik P. Microbiota and host determinants of behavioural phenotype in maternally separated mice. Nat Commun. 2015 Jul 28;6:7735. doi: 10.1038/ncomms8735. PMID 26218677
- [Result] Aizawa E, Tsuji H, Asahara T, Takahashi T, Teraishi T, Yoshida S, Ota M, Koga N, Hattori K, Kunugi H. Possible association of Bifidobacterium and Lactobacillus in the gut microbiota of patients with major depressive disorder. J Affect Disord. 2016 Sep 15;202:254-7. doi: 10.1016/j.jad.2016.05.038. Epub 2016 May 24. PMID 27288567
- [Result] Wallace CJK, Milev R. The effects of probiotics on depressive symptoms in humans: a systematic review. Ann Gen Psychiatry. 2017 Feb 20;16:14. doi: 10.1186/s12991-017-0138-2. eCollection 2017. PMID 28239408
- [Result] Kazemi A, Noorbala AA, Azam K, Eskandari MH, Djafarian K. Effect of probiotic and prebiotic vs placebo on psychological outcomes in patients with major depressive disorder: A randomized clinical trial. Clin Nutr. 2019 Apr;38(2):522-528. doi: 10.1016/j.clnu.2018.04.010. Epub 2018 Apr 24. PMID 29731182
- [Result] Akkasheh G, Kashani-Poor Z, Tajabadi-Ebrahimi M, Jafari P, Akbari H, Taghizadeh M, Memarzadeh MR, Asemi Z, Esmaillzadeh A. Clinical and metabolic response to probiotic administration in patients with major depressive disorder: A randomized, double-blind, placebo-controlled trial. Nutrition. 2016 Mar;32(3):315-20. doi: 10.1016/j.nut.2015.09.003. Epub 2015 Sep 28. PMID 26706022